CLINICAL TRIAL: NCT05412095
Title: Evaluation of the Prognostic Value of Preoperative Quadriceps and Respiratory Muscle Thickness by Ultrasound Measurement in Cardiac and Thoracic Surgery Patients: a Prospective Observational Study
Brief Title: Evaluation of the Prognostic Value of Preoperative Quadriceps and Respiratory Muscle Thickness by Ultrasound Measurement in Cardiac and Thoracic Surgery Patients
Acronym: MUSCA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BERTHOUD 2021
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery With Extracorporeal Circulation; Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiology patient: Patient requiring cardiac surgery with bypass
  Interventions: Other: Ultrasound of the abdominal wall muscles; Other: Ultrasound quadricipital; Other: Ultrasound of the diaphragm; Other: Ultrasound of the inter-costal muscles
- Pneumology patient: Patient requiring lung surgery with resection of at least one lobe
  Interventions: Other: Ultrasound of the abdominal wall muscles; Other: Ultrasound quadricipital; Other: Ultrasound of the diaphragm; Other: Ultrasound of the inter-costal muscles

INTERVENTIONS:
Other: Ultrasound of the abdominal wall muscles — the measurements will be performed during inspiration and expiration to take into account variability during the respiratory cycle. The examination is performed bilaterally and comparatively and lasts between 3 and 5 minutes.
Other: Ultrasound quadricipital — The examination is performed bilaterally and comparatively and takes between 3 and 5 minutes.
Other: Ultrasound of the diaphragm — The examination is performed bilaterally and comparatively and takes between 5 and 10 minutes.
Other: Ultrasound of the inter-costal muscles — measurements performed bilaterally on a patient in a half-sitting position at 45° and in spontaneous ventilation
Other: Ultrasound of the inter-costal muscles — In spontaneous ventilation, lying down, arms by the side of the body, palms up, head down

SUMMARY:
Cardiac and thoracic surgery are major procedures. In order to estimate the operative risk, many scores have been developed, including the Euroscore 2 in cardiac surgery. However, the Euroscore has limitations since it does not assess all the parameters that may influence postoperative complications, such as the patient's general condition or the status of his or her functional reserves.

However, it has been shown that the preoperative functional reserves have a significant impact on the patient's risk of developing postoperative complications following major surgery. In addition, there is a strong association between cardiac failure and a well-described decrease in peripheral muscle lean mass (sarcopenia) in patients older than 65 years.

Usually, a nutritional assessment is performed during the pre-anesthesia consultation. This assessment is based on clinical and biological criteria that are not totally predictive of the patient's functional reserve status.

Lean body mass (muscle) is a well-validated marker for the assessment of patients' functional reserves. However, the techniques used to date are complex and require radiation.

This study aims to use ultrasound of muscle groups (respiratory muscles - Quadriceps muscle - Diaphragm) to study the relationship between preoperative muscle mass and postoperative complications in patients over 65 years of age undergoing cardiac or thoracic surgery.

This is a prospective observational study to be conducted at the Dijon University Hospital by the cardiovascular anesthesia-intensive care department. A total of 300 patients will participate in this study, and we have planned to complete the project over a 2-year period. The participating patients (if they do not present any exclusion criteria and are not opposed to inclusion) will be included and undergo a muscle ultrasound in the cardiovascular surgery department or the thoracic and pulmonary surgery department the day before their intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient 65 years or older
* Patients who have not objected to their inclusion in the study
* Any patient requiring elective cardiac surgery, with extracorporeal circulation extracorporeal circulation OR
* Any patient requiring lung surgery with resection of at least one lobe

Exclusion Criteria:

* pneumectomy
* Person who is not affiliated to national health insurance
* Person subject to a measure of legal protection (curatorship, guardianship)
* Pregnant, parturient or breastfeeding women
* Major unable to express consent
* Persons with amputations of the proximal segment of a lower limb
* Persons suffering from a pre-existing neuromuscular pathology, tetra or paraplegia
* Person who must undergo emergency surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patient requiring cardiac or thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Onset of acute renal failure | Within 30 days after surgery
Occurrence of a respiratory complication | Within 30 days after surgery
  Occurrence of acute respiratory failure in cardiac surgery and occurrence of a severe extra-respiratory complication according to the european perioperative clinical outcome definition in pulmonary surgery
Occurrence of a cardiovascular complication | Within 30 days after surgery
Occurrence of an infectious complication | Within 30 days after surgery
Death | Within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Berthoud V, Nguyen M, Vinay J, Perrot J, Pages PB, Guinot PG, Bouhemad B. Increase in Diaphragm and Expiratory respiratory muscles thickness is not associated with postoperative pulmonary complications after thoracic surgery: a prospective ultrasound cohort study. Anaesth Crit Care Pain Med. 2025 Nov 12:101683. doi: 10.1016/j.accpm.2025.101683. Online ahead of print. PMID 41238178